CLINICAL TRIAL: NCT06170034
Title: Post-emergency Management of Patients With Transient Ischemic Attack
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Responsible Party: Sponsor
Other Study IDs: PEC AIT 84
Record Dates: First submitted 2023-11-17; First posted 2023-12-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Transient Ischemic Attack
Keywords: Emergency; Cerebral RMI; Guidelines compliance
MeSH Terms: conditions — Ischemic Attack, Transient; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TIA patients
  Interventions: Behavioral: Satisfaction questionnaire; Other: Medical care questionnaire

INTERVENTIONS:
Behavioral: Satisfaction questionnaire — Satisfaction questionnaire to assess how TIA patients feels about their medical care.
Other: Medical care questionnaire — Recording appointments and results of examinations and consultations in TIA management

SUMMARY:
A transient ischemic attack (TIA) is a momentary neurological dysfunction due to a brief cessation of blood flow to a region of the brain, resulting in typical signs of stroke (hemiplegia, aphasia, dysarthria), but whose clinical symptoms typically last less than an hour, with no visible lesion on imaging. This diagnosis remains difficult and is essentially based on the clinical judgment of the physician.

Because a TIA can be a "pre-alarm" for stroke in 20-30% of cases, it needs to be treated appropriately and as early as possible in the emergency department. Stroke rates after untreated TIA are 5% within 48 hours, 10% within one month and 20% within one year. This risk is calculated using the ABCD² score which is based on the patient's risk factors and the clinical manifestations of TIA. Patients with a score ≥ 3 should be hospitalized as soon as possible for a complete medical evaluation. However, this score has not been scientifically validated, and several specialists agree that all TIAs should be evaluated immediately. Preventing stroke is a major public health issue because it is a serious, disabling and sometimes fatal disease. Given the seriousness of the progression from TIA to stroke, the French National Authority for Health has issued a series of management recommendations. However, in practice, these guidelines remain complicated to follow and patients management may vary and be more or less effective.

Therefore, the aim of this study is to highlight the differences in how inpatients and outpatients are managed. Following these observations, solutions will be sought to make the care and management of these patients more efficient and more in line with recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Consultation in the emergency department.
* Suspected TIA diagnosed by emergency physician.
* Duration of TIA symptoms <1 hour.

Exclusion Criteria:

* Validation MRI performed prior to suspected TIA.
* Patient hospitalized for a condition other than TIA, including stroke.
* Patient referred to another hospital for further examination.
* Pregnant women.
* Patient unable to understand and answer a questionnaire.
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of TIA in the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Assess time between arrival in the emergency department for suspected TIA patients and MRI. | Baseline

SECONDARY OUTCOMES:
Time between arrival in the emergency department and MRI by departments. | Baseline
Time between arrival in the emergency department and MRI by ABCD² score. | Baseline
Percentage of patients with complete TIA management by departments. | Baseline
Hospitalization times according to care units | Baseline
Hospitalization times according to complete TIA management | Baseline
Percentage of patients with secondary event, according to complete TIA management | Baseline
Number of outpatients without complete TIA management one month after TIA. | At 1 month follow-up
Patient satisfaction with a short questionnaire | At 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yohan Fouilhe, Medical Intern, Principal Investigator — Centre Hospitalier d'Avignon, Service des urgences
Locations (1):
- Centre Hospitalier d'Avignon, Avignon, France

IPD SHARING:
Plan to Share IPD: No